CLINICAL TRIAL: NCT01860469
Title: Does Soaking Synthetic Mesh in Vancomycin Solution Reduce Mesh Infections in Open Hernia Repairs?
Brief Title: Reducing Mesh Infections in Open Hernia Repairs
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Ali Cadili, Clinical Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MeshVanco
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Patients Undergoing Open Hernia Repair; Patients Undergoing Ventral or Inguinal Hernia Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plain mesh (Active Comparator): standard practice of using plain mesh (non vancomycin-soaked) for open hernia repair
  Interventions: Procedure: plain mesh
- vancomycin-soaked mesh (Experimental): use of vancomycin-soaked mesh for open hernia repair
  Interventions: Procedure: vancomycin-soaked mesh

INTERVENTIONS:
Procedure: vancomycin-soaked mesh
  Arms: vancomycin-soaked mesh
Procedure: plain mesh
  Other Names: non vancomycin-soaked mesh
  Arms: plain mesh

SUMMARY:
Soaking meshes in a vancomycin solution just prior to their use in open hernia repairs will decrease rates of mesh infection

ELIGIBILITY:
Inclusion Criteria:

* open ventral or inguinal hernia repair

Exclusion Criteria:

* laparoscopic hernia repair
* non ventral or inguinal hernia repairs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
mesh infections | 6 months

SECONDARY OUTCOMES:
hernia recurrence | 6 months
postoperative seroma formation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Five Hills Health Region, Moose Jaw, Saskatchewan, Canada